CLINICAL TRIAL: NCT00425607
Title: An Open Label Dose Adjusted Phase II Trial of the Oral Farnesyltransferase Inhibitor (FTI) Lonafarnib (SCH66336) for Patients With Hutchinson-Gilford Progeria Syndrome (HGPS) and Progeroid Laminopathies
Brief Title: Phase II Trial of Lonafarnib (a Farnesyltransferase Inhibitor) for Progeria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Monica E. Kleinman (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor-Investigator, Monica E. Kleinman, Critical Care, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-01-007; P05009 (Other: Schering-Plough); NCT00426088 (obsolete NCT alias)
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Progeria; Hutchinson-Gilford Syndrome
Keywords: Hutchinson-Gilford Progeria Syndrome; HGPS; Progeria; FTI; Farnesyltransferase Inhibitor; Lonafarnib
MeSH Terms: conditions — Progeria | interventions — lonafarnib

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lonafarnib (Experimental): All subjects initiated oral Lonafarnib twice daily at a dose of 115mg/m2 and escalated to 150 mg/m2. Two subjects de-escalated to 115mg/m2 following toxicity.
  Interventions: Drug: Lonafarnib

INTERVENTIONS:
Drug: Lonafarnib — Lonafarnib will be taken orally, twice per day, by all patients enrolled on this study. The drug is supplied to patients in capsule form, and for patients who are unable to swallow pills, the drug may be dissolved into solution. Every patient will start lonafarnib therapy at a dose of 115mg/kg. The study allows for patients to receive a dose escalation (up to 150mg/kg) if the drug is being well-tolerated. Every patient enrolled on this study will undergo two years of lonafarnib therapy.
  Other Names: SCH66336

SUMMARY:
This is an open label dose adjusted phase II trial of the oral farnesyltransferase inhibitor (FTI) lonafarnib (SCH66336) for patients with HGPS and progeroid laminopathies.

DETAILED DESCRIPTION:
Hutchinson-Gilford Progeria Syndrome (HGPS) is a rare "premature aging" disease in which all children die at an average age of thirteen years (range 8-20 years) of severe atherosclerosis leading to strokes and heart attacks. It is a multisystem disease with objective clinical markers for disease progression. These include abnormalities in growth and body composition, bone mineral density, joint function, endocrine function, alopecia, and vascular disease. There is no effective therapy for any of the progressive and deleterious aspects of this disorder.

The gene defect causing HGPS and most progeroid laminopathies has been identified as a mutation in the gene LMNA, coding for the nuclear protein lamin A. Lamin A is normally expressed by most differentiated cells, and requires posttranslational farnesylation to incorporate into the nuclear membrane. The lamin A C-terminal peptide, including the farnesyl group, is subsequently cleaved, and mature lamin A becomes a prominent component of the nuclear scaffold just internal to the nuclear membrane, affecting nuclear structure and function.

In most cases, HGPS is a sporadic autosomal dominant disease caused by a single base alteration (henceforth designated as G608G) in the LMNA gene, which creates a cryptic splice site giving rise to an altered lamin A protein product in which 50 amino acids are deleted. The defective protein product in HGPS (henceforth progerin) lacks the cleavage site for removal of the C-terminal farnesylated peptide, and likely produces disease via dominant negative effects on the nuclear structure and function of various cell types that express lamin A. Most other progeroid laminopathies are caused by various mutations in the LMNA gene, which also subsequently creates abnormally functioning lamin A.

Lonafarnib is a farnesyltransferase inhibitor that blocks the post-translational farnesylation of prelamin A and other proteins that are targets for farnesylation. Farnesylation is essential for the function of both mutant and non-mutant lamin A proteins, including progerin. Therefore, farnesyltransferase inhibitors are ideal candidates for treatment of HGPS, which is caused by a protein (progerin) that likely depends on carrying a farnesyl group to execute its aberrant functions.

Both cell culture and mouse model studies of HGPS demonstrate improved phenotype after exposure to FTI. In vitro, exposure of HGPS skin fibroblasts and progerin-transfected HeLa cells to FTIs, including lonafarnib, prevents preprogerin from intercalating into the nuclear membrane where it normally functions, and eliminates nuclear deformity. In vivo, three Progeria-like mouse models show no appreciable signs of toxicity after FTI administration. In all three of these models, disease is significantly reduced when compared to age-matched controls after oral administration of FTI.

We propose that clinical features of HGPS can be ameliorated or reversed by blocking posttranslational farnesylation via treating patients with lonafarnib. We hypothesize that reduction of the quantity of functional progerin or, in the case of other progeroid laminopathies, other abnormal lamin proteins, will improve disease signs, symptoms and outcome. We also hypothesize that the toxicity profile of FTI inhibition using lonafarnib will be similar to that observed in children with malignant brain tumors treated with the compound.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have confirmatory mutational analysis showing G608G mutation in the lamin A gene.
* Patients with progeroid laminopathies, showing clinical signs of Progeria but with other confirmed mutations in LMNA will be eligible for therapy. This population will be analyzed separately from those with the classical mutations.
* Patients must be willing and able to come to Boston for appropriate studies and examinations approximately once every 4 months.
* Patients must have a minimum of one year of weight data available, with five data points or more, each separated by one month or more over a one year period and approval by the study team.
* APC (ANC + bands + monocytes = APC) > 1,000/ml, Platelets > 75,000/ml (transfusion independent); Hemoglobin >9g/dl.
* creatinine less than or equal to 1.5 times normal for age or GFR > 70 ml/min/1.73m2.
* bilirubin less than or equal to 1.5 x upper limit of normal for age; SGPT (ALT) < and SGOT (AST) < 5 x normal range for age.
* PT/PTT < 120% upper limit of normal OR PI approval.
* No overt renal, hepatic, pulmonary disease or immune dysfunction.
* Patients taking growth hormone when entering the study must have pretreatment weight measures while on growth hormone which are specified above. In addition, patients must remain on growth hormone treatment for the duration of the present clinical trial. Patients entering the trial not on growth hormone must remain off of growth hormone for the duration of their participation.
* Signed informed consent according to institutional guidelines must be obtained and patient must begin therapy within twenty eight (28) days.

Exclusion Criteria:

* Patient must not be receiving any other experimental drug therapy.
* Patients must not be taking medications that significantly affect the metabolism of lonafarnib.
* Subjects who have known or suspected hypersensitivity to any of the excipients included in the formulation should not be treated.
* Patients must not be pregnant or breast-feeding. Female patients of childbearing potential must have negative serum or urine pregnancy test. Male and female patients of reproductive potential must agree to use a medically accepted form of birth control while on study and up to 10 weeks after treatment. It is permissible for female patients to take oral contraceptives or other hormonal methods while receiving treatment with lonafarnib.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Kieran, MD, PhD, Study Chair — Dana-Farber Cancer Institute, Children's Hospital Boston
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Gordon LB, Kleinman ME, Miller DT, Neuberg DS, Giobbie-Hurder A, Gerhard-Herman M, Smoot LB, Gordon CM, Cleveland R, Snyder BD, Fligor B, Bishop WR, Statkevich P, Regen A, Sonis A, Riley S, Ploski C, Correia A, Quinn N, Ullrich NJ, Nazarian A, Liang MG, Huh SY, Schwartzman A, Kieran MW. Clinical trial of a farnesyltransferase inhibitor in children with Hutchinson-Gilford progeria syndrome. Proc Natl Acad Sci U S A. 2012 Oct 9;109(41):16666-71. doi: 10.1073/pnas.1202529109. Epub 2012 Sep 24. PMID 23012407
- [Result] Gordon LB, Massaro J, D'Agostino RB Sr, Campbell SE, Brazier J, Brown WT, Kleinman ME, Kieran MW; Progeria Clinical Trials Collaborative. Impact of farnesylation inhibitors on survival in Hutchinson-Gilford progeria syndrome. Circulation. 2014 Jul 1;130(1):27-34. doi: 10.1161/CIRCULATIONAHA.113.008285. Epub 2014 May 2. PMID 24795390
- [Result] Cleveland RH, Gordon LB, Kleinman ME, Miller DT, Gordon CM, Snyder BD, Nazarian A, Giobbie-Hurder A, Neuberg D, Kieran MW. A prospective study of radiographic manifestations in Hutchinson-Gilford progeria syndrome. Pediatr Radiol. 2012 Sep;42(9):1089-98. doi: 10.1007/s00247-012-2423-1. Epub 2012 Jul 1. PMID 22752073
- [Result] Ullrich NJ, Silvera VM, Campbell SE, Gordon LB. Craniofacial abnormalities in Hutchinson-Gilford progeria syndrome. AJNR Am J Neuroradiol. 2012 Sep;33(8):1512-8. doi: 10.3174/ajnr.A3088. Epub 2012 Mar 29. PMID 22460337
- [Result] Silvera VM, Gordon LB, Orbach DB, Campbell SE, Machan JT, Ullrich NJ. Imaging characteristics of cerebrovascular arteriopathy and stroke in Hutchinson-Gilford progeria syndrome. AJNR Am J Neuroradiol. 2013 May;34(5):1091-7. doi: 10.3174/ajnr.A3341. Epub 2012 Nov 22. PMID 23179651
- [Result] Ullrich NJ, Kieran MW, Miller DT, Gordon LB, Cho YJ, Silvera VM, Giobbie-Hurder A, Neuberg D, Kleinman ME. Neurologic features of Hutchinson-Gilford progeria syndrome after lonafarnib treatment. Neurology. 2013 Jul 30;81(5):427-30. doi: 10.1212/WNL.0b013e31829d85c0. Epub 2013 Jun 28. PMID 23897869
- [Derived] Suzuki M, Jeng LJB, Chefo S, Wang Y, Price D, Li X, Wang J, Li RJ, Ma L, Yang Y, Zhang X, Zheng N, Zhang K, Joseph DB, Shroff H, Doan J, Pacanowski M, Smpokou P, Donohue K, Joffe HV. FDA approval summary for lonafarnib (Zokinvy) for the treatment of Hutchinson-Gilford progeria syndrome and processing-deficient progeroid laminopathies. Genet Med. 2023 Feb;25(2):100335. doi: 10.1016/j.gim.2022.11.003. Epub 2022 Dec 12. PMID 36507973
- [Derived] Gerhard-Herman M, Smoot LB, Wake N, Kieran MW, Kleinman ME, Miller DT, Schwartzman A, Giobbie-Hurder A, Neuberg D, Gordon LB. Mechanisms of premature vascular aging in children with Hutchinson-Gilford progeria syndrome. Hypertension. 2012 Jan;59(1):92-7. doi: 10.1161/HYPERTENSIONAHA.111.180919. Epub 2011 Nov 14. PMID 22083160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 26 patients with classic HGPS from 16 countries were enrolled from May through October 2007 at Boston Children's Hospital. 2 additional patients had nonclassic mutations and are not included in the analyses.
Pre-assignment Details: One additional patient signed consent but withdrew from the protocol before receiving therapy.
Groups:
- Lonafarnib: Lonafarnib (Merck & Co., Inc.) dosing was initiated at 115 mg/m2 and was increased to 150 mg/m2 after an adjustment period of at least 4 mo. Dosage was reduced back to 115 mg/m2 for patients experiencing drug-related grade 3 or 4 toxicity and also not responding to supportive care. Once dosage was reduced, patients were permitted to increase the dose of lonafarnib. Patients received oral lonafarnib either by capsule or liquid suspension dispersed in Ora-Blend SF or Ora-Plus (Paddock Laboratories, Inc.) every 12 ± 2 h for a period of 24-29 mo.
Period: Overall Study
Arm/Group | Lonafarnib
Started | 29
Received Treatment | 28
Completed | 27
Not Completed | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The analysis population represents the 25 patients with classic HGPS who received the farnesyltransferase inhibitor lonafarnib for a minimum of 2 y. The analysis population does not include 1 patient (with prior history of strokes) who died of a stroke after 5 mo on study, or 2 additional patients who had nonclassic mutations.
Groups:
- Lonafarnib: Lonafarnib (Merck & Co., Inc.) dosing was initiated at 115 mg/m2 and was increased to 150 mg/m2 after an adjustment period of at least 4 mo. Dosage was reduced back to 115 mg/m2 fo patients experiencing drug-related grade 3 or 4 toxicity and also not responding to supportive care. Once dosage was reduced, patients were permitted to increase the dose of lonafarnib. Patients received oral lonafarnib either by capsule or liquid suspension dispersed in Ora-Blend SF or Ora-Plus (Paddock Laboratories, Inc.) every 12 ± 2 h for a period of 24-29 mo.
Arm/Group | Lonafarnib
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.0 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Successful Rate of Weight Gain
Description: Activity was assessed by determining the change in rate of weight gain over two years from baseline (determined pre-therapy for each patient).
  Primary outcome success was predefined as a 50% increase over pre-therapy in estimated annual rate of weight gain, or change from pre-therapy weight loss to statistically significant on-study weight gain.
Time Frame: Assessed at weeks 16, 32, 52, 68, 84 and 104
Population: Results are reported for the 25 patients with classic HGPS who completed at least 2y of therapy. One additional patient with a prior history of strokes died of a stroke after 5 mo on study and is not included in the analysis. Two additional patients had nonclassic mutations and are not included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Lonafarnib
Number analyzed (Participants) | 25
proportion of participants | 0.36 [0.18 to 0.58]

ADVERSE EVENTS:
Time Frame: Up to 2 years: Assessed at a minimum at weeks 16, 32, 52, 68, 84 and 104
Groups:
- Lonafarnib: Lonafarnib (Merck & Co., Inc.) dosing was initiated at 115 mg/m2 and was increased to 150 mg/m2 after an adjustment period of at least 4 mo. Dosage was reduced back to 115 mg/m2 fo patients experiencing drug-related grade 3 or 4 toxicity and also not responding to supportive care. Once dosage was reduced, patients were permitted to increase the dose of lonafarnib. Patients received oral lonafarnib either by capsule or liquid suspension dispersed in Ora-Blend SF or Ora-Plus (Paddock Laboratories, Inc.) every 12 ± 2 h for a period of 24-29 mo. Patients were monitored for liver, kidney, and hematological toxicity each month for the first 3 mo by their local physicians and every 4 mo in Boston for the duration of the study. Adverse events were monitored and recorded throughout the study.
Arm/Group | Lonafarnib
Serious Adverse Events (participants affected / at risk) | 10/28
Other Adverse Events (participants affected / at risk) | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonafarnib (N=28)
Vomiting (Gastrointestinal disorders) | 2 (2)
Stroke (Nervous system disorders) | 3 (3)
Bacterial infection (Infections and infestations) | 1 (1) — H. Pylori infection
Subdural hematoma (Nervous system disorders) | 1 (1)
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy: Sensory (Nervous system disorders) | 1 (1) — Paresthesia
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was an open label clinical trial on a very rare disease population. Patient numbers are small, though 26 participants represents a significant portion of the world's population of children with HGPS

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No